CLINICAL TRIAL: NCT06168136
Title: Effects of Medical High Protein Nutrition on the Muscle Mass in Adult ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Esam, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: protein on muscle mass in ICU
Record Dates: First submitted 2023-12-01; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Nutrient Deficiency
Keywords: muscle ultrasound; nutrition; protein diet; ICU

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Group A: included (42) patients who will receive high protein intake (target: 1.8 g protein/kg body weight /d).
  Interventions: Other: protein diet
- Control (Other): Group B: included (42) patients who will receive Standard of nutrition Care: (target: 1.2 g protein/kg body weight /d)
  Interventions: Other: Normal protein diet

INTERVENTIONS:
Other: protein diet — this group of patients will receive high protein intake (target: 1.8 g protein/kg BW/d)
  Arms: Intervention
Other: Normal protein diet — this group of patients will receive normal protein intake (target: 1.2 g protein/kg BW/d)
  Arms: Control

SUMMARY:
The use of ultrasound in clinical practice is feasible for monitoring muscle mass in critically ill patients. Assessment of muscle mass by ultrasound is clinically relevant and adds value for guiding therapeutic interventions, such as nutritional and physical therapy interventions to maintain muscle mass and promote recovery in critically ill patients.

DETAILED DESCRIPTION:
Critical illness is characterized by substantial hormone- and cytokine-mediated protein metabolism changes in various organs, leading to increased breakdown and decreased synthesis rates. Consequently, a considerable and life-threatening loss of muscle mass occurs. Medical therapeutic measures such as long-term sedation and mechanical ventilation during ICU stay can further enhance this muscle degradation (up to 2 % muscle mass per day leading to clinically relevant symptoms known as ICU-acquired weakness. Nutritional modulation, particularly of dietary amino acids, may have benefits to prevent or attenuate disease-induced muscle wasting. while there are several accurate muscle mass measurement methods and techniques [including computed tomography (CT) scan, bio-impedance analysis and ultrasound], not all are routinely feasible in clinical ICU practice. The use of ultrasound in assessing muscle mass in critically ill patients has gained much attention recently as it is non-invasive and can easily be utilized at the bedside. There are two main goals for the assessment of muscle mass: first, to assess the current muscle mass for the patient as part of (nutritional) diagnosis, and thereby risk stratification and second, to monitor the progression of muscle loss and/or recovery of muscle mass, and create opportunity to examine the effectiveness of therapeutic interventions to reduce muscle loss and/or promote muscle recovery.

ELIGIBILITY:
Inclusion Criteria:

* all critically ill-patients with Acute Physiologic Assessment and Chronic Health Evaluation II (8) (APACHE II score ) ≥ 25 and could be enterally or parenterally fed in the critical care unit of Assiut University Hospitals.

Exclusion Criteria:

* patients with malabsorption syndrome, previously diagnosed myopathies, traumatic brain injuries, intracerebral hemorrhages and cerebral ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring muscle mass changes in response to high protein intake | one year
  muscle mass using ultrasound and laboratory: titre of CK (Creatinine kinase) level.

SECONDARY OUTCOMES:
- Duration of mechanical ventilation in days. - Improvement of APACHE II score. - Duration of hospital stay in days. - Early ambulation of patients in days. - In hospital mortality. | one year
  APACHE II score is Acute Physiology and Chronic Health Evaluation II: an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Esam, Master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Wandrag L, Brett SJ, Frost GS, Bountziouka V, Hickson M. Exploration of muscle loss and metabolic state during prolonged critical illness: Implications for intervention? PLoS One. 2019 Nov 14;14(11):e0224565. doi: 10.1371/journal.pone.0224565. eCollection 2019. PMID 31725748
- [Background] Arabi YM, Al-Dorzi HM, Sadat M. Protein intake and outcome in critically ill patients. Curr Opin Clin Nutr Metab Care. 2020 Jan;23(1):51-58. doi: 10.1097/MCO.0000000000000619. PMID 31743123
- [Background] Brook MS, Wilkinson DJ, Atherton PJ. Nutrient modulation in the management of disease-induced muscle wasting: evidence from human studies. Curr Opin Clin Nutr Metab Care. 2017 Nov;20(6):433-439. doi: 10.1097/MCO.0000000000000413. PMID 28832372
- [Background] Looijaard WGPM, Molinger J, Weijs PJM. Measuring and monitoring lean body mass in critical illness. Curr Opin Crit Care. 2018 Aug;24(4):241-247. doi: 10.1097/MCC.0000000000000511. PMID 29847342
- [Background] van Ruijven IM, Stapel SN, Molinger J, Weijs PJM. Monitoring muscle mass using ultrasound: a key role in critical care. Curr Opin Crit Care. 2021 Aug 1;27(4):354-360. doi: 10.1097/MCC.0000000000000846. PMID 33973896
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Long CL, Schaffel N, Geiger JW, Schiller WR, Blakemore WS. Metabolic response to injury and illness: estimation of energy and protein needs from indirect calorimetry and nitrogen balance. JPEN J Parenter Enteral Nutr. 1979 Nov-Dec;3(6):452-6. doi: 10.1177/014860717900300609. PMID 575168